CLINICAL TRIAL: NCT07147738
Title: The Effectiveness of a Dutch School-based Prevention Program on Social-emotional Skills and Juvenile Delinquency in Children: A Randomized Controlled Trial
Brief Title: The Effectiveness of a Dutch Prevention Program on Social-emotional Skills and Juvenile Delinquency in Children
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Marit van de Mheen (Other)
Collaborators: Netherlands Institute for the Study of Crime and Law Enforcement (Unknown); VU University of Amsterdam (Other)
Responsible Party: Sponsor-Investigator, Marit van de Mheen, PhD candidate, Utrecht University
Organization: Utrecht University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1434.201.001
Record Dates: First submitted 2025-08-15; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: At Risk for Criminal Behavior

STUDY DESIGN:
Intervention Model Description: A cluster RCT will be used to determine the effectiveness of the program Incredibly Strong. Within each school, classes will be randomly assigned to either the experimental group, in which the program starts as soon as possible, or to a waitlist control group, which starts after the follow-up period (three months). Randomization to either the experimental or control group will take place using a computerized randomization in a 1:1 ratio. Classes in the waitlist control group receive the program approximately 5 months later, but still within the same school year, allowing all classes to receive the program.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): This group will participate in the program Kapot Sterk.
  Interventions: Behavioral: Kapot Sterk (translate as Incredibly Strong)
- control group (No Intervention): This group will not participate in the program. They will receive the program afterwards, once data collection is finished.

INTERVENTIONS:
Behavioral: Kapot Sterk (translate as Incredibly Strong) — The program consists of five lessons of approximately 60 minutes long, delivered over a period of four to eight weeks. The lessons are facilitated by trained pedagogical staff (e.g., youth workers), while the school's own teachers are always present during the sessions. Lessons include active learning strategies such as role-playing, group discussions, and reflection exercises, often based on realistic and recognizable scenarios. The program focuses on strengthening key social-emotional skills, such as self-esteem, self-control, and resistance to peer pressure.
  Arms: experimental group

SUMMARY:
The purpose of this study is to investigate whether the prevention program Kapot Sterk is effective.

DETAILED DESCRIPTION:
Given the growing concerns about youth's involvement in criminal behavior, there is a strong need for effective interventions to prevent it. However, knowledge about the effectiveness of prevention programs for juveniles is currently lacking. Incredibly Strong (translate as Kapot Sterk) is a prevention program designed to improve self-esteem, self-control, and resistance to peer pressure among pupils in elementary schools. By enhancing these social-emotional skills, the program ultimately aims to reduce youths' vulnerability to recruitment and involvement in criminal activities. The effects of Incredibly Strong on juvenile delinquency and other life domains are investigated, using a randomized controlled trial (RCT).

ELIGIBILITY:
Inclusion Criteria:

Every pupil who meets the inclusion criteria for the intervention program can participate in the study. The program is for pupils in their last or second-to-last year of elementary school.

* Participants are 10-13 years old.
* Participants attend school.

Exclusion Criteria:

- Participants are younger than 10 years old or older than 13 years old.

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Estimated)
Dates: Start 2024-11-20 (Actual); Primary Completion 2025-09-26 (Estimated); Study Completion 2025-09-26 (Estimated)

PRIMARY OUTCOMES:
Self-esteem | baseline (T0), immediately after the program ended for the intervention group (or after the waiting period for the control group) (T1), and at 3 months post-program (T2).
  will be measured using an instrument based on items from the Dutch version of the Rosenberg Self-Esteem Scale (RSES), developed for a study with children aged 8-12 years. The instrument contains five items (e.g., "I think positively about myself"), rated on a 3-point scale ranging from 1 (not true) to 3 (definitely true). Higher scores reflect greater self-esteem.
Self-control | baseline (T0), immediately after the program ended for the intervention group (or after the waiting period for the control group) (T1), and at 3 months post-program (T2).
  will be measured using five items based on the Brief Self-Control Scale (Tangney et al., 2004) (e.g., "I am good at saying no to things that are hard to resist"). Items are rated on a 5-point Likert scale ranging from 1 (strongly disagree) to 5 (strongly agree). Items 3 and 4 will be reverse coded so that higher scores reflect higher self-control.
Peer pressure | baseline (T0), immediately after the program ended for the intervention group (or after the waiting period for the control group) (T1), and at 3 months post-program (T2).
  will be measured using ten items based on the Peer Pressure Scale (Sullivan, 2006). The original items have been translated into Dutch and adapted to reflect minor offenses typically committed by juveniles (e.g., "I feel pressure from my friends to steal something from a shop"). Items are rated on a 5-point Likert scale ranging from 1 (absolutely never) to 5 (very often). Higher scores indicate greater levels of experienced peer pressure.

SECONDARY OUTCOMES:
Externalizing behavior | baseline (T0) and at 3 months post-program (T2).
  will be measured using the externalizing behavior and delinquency subscales of the Youth Self-Report (YSR) (Verhulst & Van der Ende, 1992). The instrument focuses on various externalizing behaviors, including aggression and delinquent behavior. The YSR includes items such as "I fight a lot", which are rated on a 3-point Likert scale ranging from 0 (never) to 2 (often). Higher scores on the YSR externalizing subscale indicate greater levels of externalizing behavior.
Perceived social support from parents, friends, and significant others | baseline (T0), immediately after the program ended for the intervention group (or after the waiting period for the control group) (T1), and at 3 months post-program (T2).
  will be measured using the 12-item Multidimensional Scale of Perceived Social Support (MSPSS) (Zimet et al., 1990). Participants rate statements such as "I have a special person who is a real source of comfort to me" and "I can talk about my problems with my family" on a 5-point Likert scale (1 = very strongly disagree to 5 = very strongly agree). Higher scores indicate greater levels of experienced support.
Knowledge of youth work | baseline (T0), immediately after the program ended for the intervention group (or after the waiting period for the control group) (T1), and at 3 months post-program (T2).
  will be assessed using four questions. Participants are first asked, "How well do you know what youth work is?" Those who respond with "well" or "a little" are then prompted to describe, in their own words, what youth workers do. A similar procedure is followed for the question "How well do you know where to find youth workers?" Participants who indicate some level of knowledge are asked to specify where youth workers can be found.

OTHER OUTCOMES:
Demographic, personal, socioeconomic, and family background | Baseline (T0)
  will be assessed through a questionnaire covering demographic information, including age, gender, ethnic identity, family composition, and financial situation (e.g., "Do you worry whether there is enough money at home?").
Parent-child relationship | baseline (T0) and at 3 months post-program (T2).
  will be assessed using statements based on the Parental Monitoring Questionnaire (Stattin & Kerr, 2000) containing three subscales: parental control, parental solicitation, and parental disclosure. Parental control contains five item, indicating the extent to which parents seek to regulate their child's behavior by requiring permission for leisure activities. Parental solicitation (five items) captures the degree to which parents proactively seek information about their child's leisure activities. Parental disclosure (5 items) reflects how openly juveniles voluntarily share such information with their parents. All items are rated on a 5-point Likert scale 1 (never) to 5 (always). Parental responsivity will be assessed using the eight-item Responsivity subscale of the Nijmegen Parenting Questionnaire (Gerris, 1993). Items are rated on a 6-point Likert scale ranging from 1 (strongly disagree) to 6 (strongly agree).
Presence of Deviant peers | baseline (T0) and at 3 months post-program (T2).
  will be measured using the Deviant Peers Scale from the Basic Questionnaire on Peer Relationships (Weerman & Smeenk, 2005). The five -items questionnaire assesses the extent to which juveniles have deviant friends. (e.g., ''How many of your friends have robbed someone by threatening with a weapon or violence, or by using violence?''). Responses are given on a four-point scale (none, some, most, all). Internal consistency in previous studies was high. Higher scores on this scale indicate that juveniles have more deviant friends.
Problems and help-seeking | baseline (T0) and at 3 months post-program (T2).
  will be measured using a short questionnaire that has also been used in the study of Tollenaar and colleagues (Tollenaar et al., 2024). This questionnaire asks about various issues pupils may have experienced in the past six months (e.g., family problems, financial problems, or mental health issues). Respondents can indicate whether they have had any of these problems and, if so, whether they sought help and from whom (e.g., social worker, youth services, school mentor, or parents). Responses are given as yes/no options for each category, and additional open-ended fields allow participants to specify other sources of help or problems they experienced.
School performance | baseline (T0) and at 3 months post-program (T2).
  will be measured using an adapted version the Family, Friends, and Self (FSS) questionnaire (Simpson & McBride, 1992). The questionnaire contains five items (e.g., "How did your schoolwork go last week?"). Responses are given on a five-point scale ranging from 1 (really bad) to 5 (really good), with higher scores indicating better school performance. The internal consistency is good (α = .79) (Duari & Mohapatra, 2021; Simpson & McBride, 1992). Participants are also asked whom they can ask for help with their homework and whether they skip school.
Leisure time activities | baseline (T0) and at 3 months post-program (T2).
  will be assessed using a questionnaire based on the Dutch Monitor of Self-Reported Delinquency (Tollenaar et al., 2024). Participants answered two questions about where they usually spend their time after school on weekdays (Monday to Thursday) and during the weekend (Friday to Sunday). Eleven response options were provided, allowing multiple answers. Examples include going out with parents; attending a sports club; being at friends' homes; hanging out on the street with friends; or never going out/mostly staying at home.

CONTACTS AND LOCATIONS:
Overall Officials: Jessica J Asscher, PhD., Principal Investigator — Utrecht University
Locations (1):
- Utrecht University, Utrecht, Netherlands

IPD SHARING:
Plan to Share IPD: Yes
The data can be shared in anonymized form upon request.
Supporting Information: Study Protocol
Time Frame: The data will become available after the completion of the program and data collection.